CLINICAL TRIAL: NCT06273917
Title: Deprescribing Potentially Inappropriate Medications in the Emergency Department for Persons Living With Dementia
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Scott Dresden, Dr. Scott Dresden, Northwestern University Feinberg School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: FY23_Pilot2_Dresden
Record Dates: First submitted 2024-02-05; First posted 2024-02-23 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Dementia
Keywords: Depresribing Medication
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRIDE Patients (Experimental): Community-dwelling adults (age 18+) in the ED with prior outpatient visits within the NM system and a history of dementia or mild cognitive impairment recorded in the NM EHR will be eligible for inclusion. We will include 290 patients across 3 sites to have medication reconciliation conducted by the clinical pharmacist. Patients who were previously prescribed CNS PIMs will have deprescribing recommendations communicated by the clinical pharmacist to the outpatient prescriber.
  Interventions: Other: PRIDE

INTERVENTIONS:
Other: PRIDE — Pharmacists present in the ED will perform medication reconciliation for eligible patients. This will be done to demonstrate the feasibility of the PRIDE intervention in the ED for patients with ADRD and MCI. Patients eligible for medication reconciliation will be enrolled in Aim 2 of the study.
  Outpatient prescribers of these patients who are discharged from the ED will be contacted by the ED pharmacist on the date of ED discharge and will receive a medication report including fill data 90-100 days after the ED visit.
  At the completion of the study, the outpatient clinicians will also receive a questionnaire about the acceptability of the PRIDE program including the Acceptability of Intervention Measure to complete electronically.

SUMMARY:
Aim 1: To demonstrate the feasibility by determining proportion of completed medication reconciliation, Central Nervous System active Potentially Inappropriate Medication (CNS PIM) use among patients with Alzheimer's Disease and Related Dementias (ADRD) and Mild Cognitive Impairment (MCI) in the emergency department (ED), and communication between ED clinical pharmacists and outpatient prescribers.

Aim 2: To demonstrate the feasibility of collecting the primary and secondary outcomes for a subsequent study. The future primary outcome will be reduction in CNS PIMs 90 days after an ED visit. Secondary outcomes will include outpatient follow-up, repeat ED visits, and hospitalizations during the 90 days following an ED visit.

Aim 3: To demonstrate the acceptability of the PRIDE intervention to outpatient clinicians using the Acceptability of Intervention Measure and qualitative analysis of responses.

DETAILED DESCRIPTION:
This is an embedded pragmatic clinical trial (ePCT) of the Pharmacist Reconciliation of Inappropriate medications and Deprescribing in the Emergency department (PRIDE) intervention which will be implemented as standard care for all community-dwelling adults (age 18+) in the ED with prior outpatient visits within the Northwestern Medicine (NM) healthcare system who have been diagnosed with Alzheimer's Disease and Related Dementias (ADRD) or Mild Cognitive Impairment (MCI) as clinical pharmacist availability allows. The PRIDE program did not exist prior to the initiation of this study. PRIDE is in the process of being implemented at all three hospitals and will continue beyond the end of the research study.

This study will take place at 3 hospital emergency departments within the Northwestern Medicine (NM) Healthcare System. Community-dwelling adults (age 18+) in the ED with prior outpatient visits within the NM system and a history of dementia or mild cognitive impairment recorded in the NM EHR will be eligible for the study.

The primary outcome is the number and percent of patients taking central nervous system potentially inappropriate medications (CNS PIMs) who have documented communication of pharmacist's recommendations for deprescribing on the day of the ED visit. The key secondary outcome is the number and percent of patients with ADRD or MCI in the ED who have documented medication reconciliation by the clinical pharmacist on the day of the ED visit.

Pharmacists present in the ED will perform medication reconciliation for eligible patients. This will be done to demonstrate the feasibility of the PRIDE intervention in the ED for patients with ADRD and MCI. Patients eligible for medication reconciliation will be enrolled in Aim 2 of the study.

Outpatient prescribers of these patients who are discharged from the ED will be contacted by the ED pharmacist on the date of ED discharge and will receive a medication report including fill data 90-100 days after the ED visit.

At the completion of the study, the outpatient clinicians will also receive a questionnaire about the acceptability of the PRIDE program including the Acceptability of Intervention Measure to complete electronically.

Community-dwelling adults (age 18+) in the ED with prior outpatient visits within the NM system and a history of dementia or mild cognitive impairment recorded in the NM EHR will be eligible for inclusion. We will include 290 patients across 3 sites to have medication reconciliation conducted by the clinical pharmacist. Patients who were previously prescribed CNS PIMs will have deprescribing recommendations communicated by the clinical pharmacist to the outpatient prescriber.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling
* 18 years of age or older
* History of dementia or mild cognitive impairment in the problem list in the NM EHR. A history of mild cognitive impairment will be identified using the ICD-10 code G31.84 (mild cognitive impairment) or ICD-10 codes suggestive of ADRD as described in the Bynum-standard algorithm: F01.50-F01.51 (vascular dementia), F02.80-F02.81 (dementia), F03.90-F03.91 (unspecified dementia), F04 (amnestic disorder), G30.0/30.1/30.8/G30.9 (Alzheimer's disease), G31.01 (Pick's disease), G31.09 (frontotemporal dementia), G31.83 (dementia with Lewy bodies), G31.1 (senile degeneration), G31.2 (degeneration of nervous system), R41.81 (age-related cognitive decline).
* Able to participate in medication reconciliation as determined by the pharmacist per usual care OR a care partner with knowledge of the patient's current medications is present in the ED or is available by phone.
* Has had prior outpatient care performed at Northwestern Medicine location(s)
* Arrives to the emergency department between 7am and 7pm, Monday-Friday

Exclusion Criteria:

* Emergency Severity Index (ESI) of 1 (critical)
* ICU consult placed in the ED
* Reside in nursing facility or assisted living facility

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Pharmacist communication of deprescribing recommendation | 24 hours
  This will be determined if the ED pharmacist sends an electronic message through the EHR to the outpatient prescriber with de-prescribing recommendations for patients who are taking CNS PIMs. This will be performed on Day 0 in the Emergency Department.

SECONDARY OUTCOMES:
Medication reconciliation | 24 hours
  This will be determined if the ED pharmacist enters a medication reconciliation document into the EHR. This will occur on Day 0 in the ED.
Medication supply of CNS PIMs | 90 days
  this will be determined through outpatient pharmacy records at day 90. Medication supply will be calculated using dose, frequency, and quantity data through SureScripts.
Outpatient follow up | 90 days
  the number and frequency of outpatient visits to the outpatient prescriber who received the deprescribing recommendation from day 1-90 as determined through the EHR after day 90.
Repeat Emergency Department visits | 90 days
  any ED visit which occurs within the Northwestern Medicine system from day 1-90 as determined through the EHR after day 90.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Dresden, Dr., Principal Investigator — Northwestern University- Department of Emergency Medicine
Locations (3):
- United States (3):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Northwestern Medicine Palos Hospital, Palos Heights, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hebert LE, Weuve J, Scherr PA, Evans DA. Alzheimer disease in the United States (2010-2050) estimated using the 2010 census. Neurology. 2013 May 7;80(19):1778-83. doi: 10.1212/WNL.0b013e31828726f5. Epub 2013 Feb 6. PMID 23390181
- [Background] Hunt LJ, Coombs LA, Stephens CE. Emergency Department Use by Community-Dwelling Individuals With Dementia in the United States: An Integrative Review. J Gerontol Nurs. 2018 Mar 1;44(3):23-30. doi: 10.3928/00989134-20171206-01. Epub 2018 Jan 23. PMID 29355877
- [Background] Kent T, Lesser A, Israni J, Hwang U, Carpenter C, Ko KJ. 30-Day Emergency Department Revisit Rates among Older Adults with Documented Dementia. J Am Geriatr Soc. 2019 Nov;67(11):2254-2259. doi: 10.1111/jgs.16114. Epub 2019 Aug 12. PMID 31403717
- [Background] LaMantia MA, Stump TE, Messina FC, Miller DK, Callahan CM. Emergency Department Use Among Older Adults With Dementia. Alzheimer Dis Assoc Disord. 2016 Jan-Mar;30(1):35-40. doi: 10.1097/WAD.0000000000000118. PMID 26523710
- [Background] Han JH, Wilber ST. Altered mental status in older patients in the emergency department. Clin Geriatr Med. 2013 Feb;29(1):101-36. doi: 10.1016/j.cger.2012.09.005. PMID 23177603
- [Background] Carpenter CR, Bromley M, Caterino JM, Chun A, Gerson LW, Greenspan J, Hwang U, John DP, Lyons WL, Platts-Mills TF, Mortensen B, Ragsdale L, Rosenberg M, Wilber S; ACEP Geriatric Emergency Medicine Section; American Geriatrics Society; Emergency Nurses Association; Society for Academic Emergency Medicine Academy of Geriatric Emergency Medicine. Optimal older adult emergency care: introducing multidisciplinary geriatric emergency department guidelines from the American College of Emergency Physicians, American Geriatrics Society, Emergency Nurses Association, and Society for Academic Emergency Medicine. J Am Geriatr Soc. 2014 Jul;62(7):1360-3. doi: 10.1111/jgs.12883. Epub 2014 Jun 2. PMID 24890806
- [Background] Gettel CJ, Falvey JR, Gifford A, Hoang L, Christensen LA, Hwang U, Shah MN; GEAR 2.0-ADC Network. Emergency Department Care Transitions for Patients With Cognitive Impairment: A Scoping Review. J Am Med Dir Assoc. 2022 Aug;23(8):1313.e1-1313.e13. doi: 10.1016/j.jamda.2022.01.076. Epub 2022 Mar 2. PMID 35247358
- [Background] Southerland LT, Lo AX, Biese K, Arendts G, Banerjee J, Hwang U, Dresden S, Argento V, Kennedy M, Shenvi CL, Carpenter CR. Concepts in Practice: Geriatric Emergency Departments. Ann Emerg Med. 2020 Feb;75(2):162-170. doi: 10.1016/j.annemergmed.2019.08.430. Epub 2019 Nov 13. PMID 31732374
- [Background] Dresden SM, Hwang U, Garrido MM, Sze J, Kang R, Vargas-Torres C, Courtney DM, Loo G, Rosenberg M, Richardson L. Geriatric Emergency Department Innovations: The Impact of Transitional Care Nurses on 30-day Readmissions for Older Adults. Acad Emerg Med. 2020 Jan;27(1):43-53. doi: 10.1111/acem.13880. Epub 2019 Dec 1. PMID 31663245
- [Background] Hwang U, Dresden SM, Vargas-Torres C, Kang R, Garrido MM, Loo G, Sze J, Cruz D, Richardson LD, Adams J, Aldeen A, Baumlin KM, Courtney DM, Gravenor S, Grudzen CR, Nimo G, Zhu CW; Geriatric Emergency Department Innovations in Care Through Workforce, Informatics, and Structural Enhancement (GEDI WISE) Investigators. Association of a Geriatric Emergency Department Innovation Program With Cost Outcomes Among Medicare Beneficiaries. JAMA Netw Open. 2021 Mar 1;4(3):e2037334. doi: 10.1001/jamanetworkopen.2020.37334. PMID 33646311
- [Background] Hwang U, Dresden SM, Rosenberg MS, Garrido MM, Loo G, Sze J, Gravenor S, Courtney DM, Kang R, Zhu CW, Vargas-Torres C, Grudzen CR, Richardson LD; GEDI WISE Investigators. Geriatric Emergency Department Innovations: Transitional Care Nurses and Hospital Use. J Am Geriatr Soc. 2018 Mar;66(3):459-466. doi: 10.1111/jgs.15235. Epub 2018 Jan 10. PMID 29318583
- [Background] Martinez AI, Abner EL, Jicha GA, Rigsby DN, Eckmann LC, Huffmyer MJ, Moga DC. One-Year Evaluation of a Targeted Medication Therapy Management Intervention for Older Adults. J Manag Care Spec Pharm. 2020 Apr;26(4):520-528. doi: 10.18553/jmcp.2020.26.4.520. PMID 32223601
- [Background] Wilchesky M, Mueller G, Morin M, Marcotte M, Voyer P, Aubin M, Carmichael PH, Champoux N, Monette J, Giguere A, Durand P, Verreault R, Arcand M, Kroger E. The OptimaMed intervention to reduce inappropriate medications in nursing home residents with severe dementia: results from a quasi-experimental feasibility pilot study. BMC Geriatr. 2018 Sep 4;18(1):204. doi: 10.1186/s12877-018-0895-z. PMID 30180821
- [Background] Harrison SL, Cations M, Jessop T, Hilmer SN, Sawan M, Brodaty H. Approaches to Deprescribing Psychotropic Medications for Changed Behaviours in Long-Term Care Residents Living with Dementia. Drugs Aging. 2019 Feb;36(2):125-136. doi: 10.1007/s40266-018-0623-6. PMID 30535930
- [Background] Bayliss EA, Shetterly SM, Drace ML, Norton JD, Maiyani M, Gleason KS, Sawyer JK, Weffald LA, Green AR, Reeve E, Maciejewski ML, Sheehan OC, Wolff JL, Kraus C, Boyd CM. Deprescribing Education vs Usual Care for Patients With Cognitive Impairment and Primary Care Clinicians: The OPTIMIZE Pragmatic Cluster Randomized Trial. JAMA Intern Med. 2022 May 1;182(5):534-542. doi: 10.1001/jamainternmed.2022.0502. PMID 35343999
- [Background] Houlind MB, Andersen AL, Treldal C, Jorgensen LM, Kannegaard PN, Castillo LS, Christensen LD, Tavenier J, Rasmussen LJH, Ankarfeldt MZ, Andersen O, Petersen J. A Collaborative Medication Review Including Deprescribing for Older Patients in an Emergency Department: A Longitudinal Feasibility Study. J Clin Med. 2020 Jan 27;9(2):348. doi: 10.3390/jcm9020348. PMID 32012721
- [Background] McCarthy EP, Chang CH, Tilton N, Kabeto MU, Langa KM, Bynum JPW. Validation of Claims Algorithms to Identify Alzheimer's Disease and Related Dementias. J Gerontol A Biol Sci Med Sci. 2022 Jun 1;77(6):1261-1271. doi: 10.1093/gerona/glab373. PMID 34919686
- [Background] Allore HG, Gnjidic D, Skanderson M, Han L. Association Between Potentially Inappropriate Medications and 30-Day Post-Hospital Discharge Outcomes in US Veterans. Ann Pharmacother. 2022 Mar;56(3):256-263. doi: 10.1177/10600280211032072. Epub 2021 Jul 20. PMID 34282638
- [Background] By the 2019 American Geriatrics Society Beers Criteria(R) Update Expert Panel. American Geriatrics Society 2019 Updated AGS Beers Criteria(R) for Potentially Inappropriate Medication Use in Older Adults. J Am Geriatr Soc. 2019 Apr;67(4):674-694. doi: 10.1111/jgs.15767. Epub 2019 Jan 29. PMID 30693946
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459